CLINICAL TRIAL: NCT06033079
Title: Improving CarE for Community Acquired Pneumonia 1 (ICE-CAP1): Prognostic Decision Support
Brief Title: Improving CarE for Community Acquired Pneumonia 1 (ICE-CAP2)
Acronym: ICE-CAP2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); University of Pittsburgh Medical Center (Other)
Responsible Party: Principal Investigator, Derek Williams, Associate Professor of Pediatrics, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R01AI125642pt2; R01AI125642 (NIH)
Record Dates: First submitted 2023-08-23; First posted 2023-09-13 (Actual); Results first posted 2023-12-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Pneumonia Childhood

STUDY DESIGN:
Intervention Model Description: We will conduct a randomized controlled trial comparing our prognostic tool (intervention arm) to usual care (control arm) over a period of 24 months. Randomization will occur at the patient level. Allocation to intervention or control will be based on medical record number (even vs. odd) or similar strategy and will be assigned automatically once a provider confirms the diagnosis of pneumonia. Importantly, all standard of care treatment options will be available and decision-making will not be restricted in any way in either group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CDS Intervention (Experimental): The prognostic decision support application will be provided to those randomized to the intervention arm. Due to the nature of the intervention, blinding of treating providers will not be possible. All children will receive usual care and all treatment decisions will be made by the clinical providers and will not be restricted or altered in any way.
  Interventions: Behavioral: Clinical Decision Support
- Control (No Intervention): No experimental decision support will be provided to those randomized to the control arm. All children will receive usual care and treatment will not be restricted or altered in any way by the study.

INTERVENTIONS:
Behavioral: Clinical Decision Support — For enrolled subjects assigned to the decision support arm, providers will receive prognostic information derived using our previously validated and best performing model. The decision support application will automatically calculate predicted risk for moderate (intensive care) and severe (respiratory failure or shock) outcomes using the parameters derived from the prognostic tool's regression equation. Outcome probabilities will be integrated into the decision support application and displayed within the EHR.
  Arms: CDS Intervention

SUMMARY:
Children with pneumonia presenting to the emergency department at Monroe Carell Jr. Children's Hospital at Vanderbilt or Children's Hospital of Pittsburgh will be potentially eligible for study. During intervention periods, providers caring for enrolled children will be presented with a detailed decision support strategy that emphasizes management in accordance with national guideline recommendations. The anticipated study duration is 24 months and, as this study does not include direct contact with enrolled subjects, there is no anticipated follow up.

DETAILED DESCRIPTION:
Pneumonia is the most common serious infection in childhood. In the United States (US), pneumonia accounts for 1-4% of all emergency department (ED) visits in children (3-28 per 1,000 US children per year) and ranks among the top 3 reasons for pediatric hospitalization with >100,000 hospitalizations per year (15-22 per 100,000 US children per year). Pneumonia also accounts for more days of antibiotic use in US children's hospitals than any other condition.

Emergency care for childhood pneumonia, including hospitalization rates, varies widely across the nation. A study examining hospital admission rates at 35 US children's hospitals from 2009-12 showed marked differences in severity-adjusted pneumonia hospital admission rates (median 31%; range 19-69%). Provider preferences and inaccurate risk perceptions contribute to these differences in hospitalization rates. Within the Intermountain Healthcare System in Utah, Dean et al. exposed large differences in admission rates (range 38-79%) among 18 individual ED providers providing care for >2,000 adults with pneumonia. Differences were not explained by patient characteristics or illness severity and higher rates of hospitalization did not reduce hospital readmissions or mortality. In another multicenter study of 472 adults with pneumonia at <4% risk of 30-day mortality estimated using objective severity scores, providers overestimated the risk of mortality in 5% of outpatients (range across institutions 0-12%) and 41% of inpatients (range across institutions 36-48%). These studies suggest that risk perceptions are often inaccurate, and potentially lead to unnecessary or prolonged hospitalizations and intensive therapies. Similar studies have not been performed in children because no valid prognostic tools exist to reliably predict pediatric pneumonia severity.

ELIGIBILITY:
Inclusion Criteria:

1. Six months to <18 years of age
2. Radiographic evidence of pneumonia in ED
3. Provider-confirmed diagnosis of pneumonia

Exclusion Criteria:

1. Children with tracheostomy, cystic fibrosis, immunosuppression
2. Inter-hospital transfers
3. Hospitalization within preceding 7 days
4. Previously enrolled within preceding 28 days
5. Provider preference for any reason

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 536 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Derek J Williams, MD, MPH, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Monroe Carell Jr. Children's Hospital - Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Williams DJ, Nian H, Suresh S, Slagle J, Gradwohl S, Johnson J, Stassun J, Reale C, Just SL, Rixe NS, Beebe R, Arnold DH, Turer RW, Antoon JW, Sartori LF, Freundlich RE, Grijalva CG, Smith JC, Weitkamp AO, Weinger MB, Zhu Y, Martin JM. Prognostic clinical decision support for pneumonia in the emergency department: A randomized trial. J Hosp Med. 2024 Sep;19(9):802-811. doi: 10.1002/jhm.13391. Epub 2024 May 26. PMID 38797872

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | CDS Intervention
Started | 269 | 267
Completed | 269 | 267
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | CDS Intervention | Total
Number analyzed (Participants) | 269 | 267 | 536
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 4.4 [2.1 to 7.0] | 4.3 [2.1 to 7.2] | 4.4 [2.1 to 7.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 126 | 141 | 267
  Male | 143 | 126 | 269
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 184 | 177 | 361
  Black | 36 | 50 | 86
  Asian | 4 | 2 | 6
  Other | 15 | 7 | 22
  Unknown | 30 | 31 | 61
Comorbidity [Count of Participants; unit: Participants] — Population: Data for this measure not available for all patients.
  Participants
    number analyzed (Participants) | 256 | 240 | 496
    Non-chronic | 150 | 132 | 282
    Non-complex chronic | 26 | 25 | 51
    Complex chronic | 80 | 83 | 163
Insurance [Count of Participants; unit: Participants]
  Public | 153 | 142 | 295
  Private | 95 | 101 | 196
  Multiple | 16 | 20 | 36
  None | 5 | 4 | 9
Triage temperature [Median (Inter-Quartile Range); unit: degrees Celsius] | 37.5 [36.9 to 38.2] | 37.2 [36.8 to 38.08] | 37.3 [36.8 to 38.1]
Triage heart rate [Median (Inter-Quartile Range); unit: beats per minute] | 138.5 [121.0 to 154.0] | 135.0 [117.0 to 155.0] | 136.0 [118.0 to 155.0]
Triage respiratory rate [Median (Inter-Quartile Range); unit: respirations per minute] | 30.0 [24.0 to 40.0] | 32.0 [24.0 to 40.5] | 31.0 [24.0 to 40.0]
Triage systolic blood pressure [Median (Inter-Quartile Range); unit: mmHg] | 108.0 [99.0 to 117.0] | 108.0 [100.0 to 117.0] | 108.0 [100.0 to 117.0]
SpO2:FiO2 ratio [Median (Inter-Quartile Range); unit: ratio] — Population: Data for this measure not available for all patients.
  ratio
    number analyzed (Participants) | 220 | 227 | 447
    (all) | 457.1 [442.9 to 466.7] | 457.1 [447.6 to 466.7] | 457.1 [447.6 to 466.7]

OUTCOME MEASURES:

1. Primary Outcome: Inappropriate Disposition
Description: Number of participants who were disposed from the ED and experienced a change in level of care within 24 hours unless objective criteria present. Appropriate dispositions were defined as follows.
  1. Disposition: Discharged to home, Appropriate if no subsequent hospitalization within 24h
  2. Disposition: Inpatient Ward, Appropriate if hospital length of stay (LOS) ≥ 24h OR hospital LOS < 24h with objective criteria for admission present (eg, need for supplemental oxygen) PLUS no transfer to intensive care (ICU) within 24h
  3. Disposition: ICU, ICU LOS ≥ 24h OR ICU LOS < 24h with objective criteria for ICU admission present (eg, respiratory failure)
  Encounters NOT meeting these criteria were defined as Inappropriate.
Time Frame: 24 Hours
Measure: Count of Participants; unit: Participants
Arm/Group | Control | CDS Intervention
Number analyzed (Participants) | 269 | 267
Participants | 7 | 6
Statistical Analysis 1: Comparison: Control vs CDS Intervention; Test type: Superiority; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.32 to 2.95]

2. Secondary Outcome: Overall Site-of-care Disposition
Description: This outcome reports the total number of participants who were initially discharged from the ED, admitted to the inpatient ward, or admitted to the ICU.
Time Frame: ED Disposition
Measure: Count of Participants; unit: Participants
Arm/Group | Control | CDS Intervention
Number analyzed (Participants) | 269 | 267
Participants
  ED | 107 | 109
  Inpatient | 113 | 96
  ICU | 49 | 62
Statistical Analysis 1: Comparison: Control vs CDS Intervention; Test type: Superiority; p = 0.233, Fisher Exact

3. Secondary Outcome: ED Revisits (72 Hours)
Description: This outcome reports the number of participants who presented to the ED for care within 72 hours of the index discharge.
Time Frame: 72 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Control | CDS Intervention
Number analyzed (Participants) | 269 | 267
Participants | 10 | 6
Statistical Analysis 1: Comparison: Control vs CDS Intervention; Test type: Superiority; Odds Ratio (OR) = 0.86, 95% CI 2-sided [0.30 to 2.37]

4. Secondary Outcome: ED Revisits (7 Days)
Description: This outcome reports the number of participants who presented to the ED for care within 7 days of the index discharge.
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Control | CDS Intervention
Number analyzed (Participants) | 269 | 267
Participants | 15 | 9
Statistical Analysis 1: Comparison: Control vs CDS Intervention; Test type: Superiority; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.32 to 1.82]

5. Secondary Outcome: Rehospitalizations (72 Hours)
Description: This outcome reports the number of participants who were readmitted to the hospital for pneumonia-related illness within 72 hours of the index discharge.
Time Frame: 72 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Control | CDS Intervention
Number analyzed (Participants) | 269 | 267
Participants | 2 | 9
Statistical Analysis 1: Comparison: Control vs CDS Intervention; Test type: Superiority; Odds Ratio (OR) = 1.42, 95% CI 2-sided [0.34 to 7.51]

6. Secondary Outcome: Rehospitalizations (7 Days)
Description: This outcome reports the number of participants who were readmitted to the hospital for pneumonia-related illness within 7 days of the index discharge.
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Control | CDS Intervention
Number analyzed (Participants) | 269 | 267
Participants | 8 | 5
Statistical Analysis 1: Comparison: Control vs CDS Intervention; Test type: Superiority; Hazard Ratio (HR) = 0.46, 95% CI 2-sided [0.13 to 1.42]

7. Other Pre Specified Outcome: Death
Description: This outcome reports the number of participants who died as a result of their pneumonia-related illness within 30 days discharge from the index encounter.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Control | CDS Intervention
Number analyzed (Participants) | 269 | 267
Participants | 3 | 4
Statistical Analysis 1: Comparison: Control vs CDS Intervention; Test type: Superiority; Odds Ratio (OR) = 1.72, 95% CI 2-sided [0.41 to 7.90]

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Control | CDS Intervention
All-Cause Mortality (participants affected / at risk) | 3/269 | 4/267
Serious Adverse Events (participants affected / at risk) | 0/269 | 0/267
Other Adverse Events (participants affected / at risk) | 0/269 | 0/267

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-10-26): https://cdn.clinicaltrials.gov/large-docs/79/NCT06033079/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-26): https://cdn.clinicaltrials.gov/large-docs/79/NCT06033079/SAP_001.pdf